CLINICAL TRIAL: NCT02954302
Title: Proximal Roux-en-y Gastrojejunal Anastomosis on Delayed Gastric Emptying After Pylorus-resecting Pancreaticoduodenectomy: A Randomized Controlled Trial
Brief Title: Proximal Roux-en-y Gastrojejunal Anastomosis on Delayed Gastric Emptying After Pylorus-resecting Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: LanZhou University (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAHXMU-2016-04
Record Dates: First submitted 2016-09-07; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Cancer; Bile Duct Cancer; Duodenal Cancer
Keywords: Delayed gastric emptying; pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms; Duodenal Neoplasms; Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PrPD with RGA (Experimental): Patients who will undergo PrPD with proximal Roux-en-y gastrojejunal anastomosis.
  Interventions: Procedure: PrPD with proximal Roux-en-y gastrojejunal anastomosis
- conventional PrPD (Experimental): Patients who will undergo conventional PrPD.
  Interventions: Procedure: conventional PrPD

INTERVENTIONS:
Procedure: PrPD with proximal Roux-en-y gastrojejunal anastomosis — the distal antrum was divided about 1 to 2 cm proximal to the pylorus ring, preserving more than 95% of the stomach. The proximal jejunum was divided approximately 2 to 4 cm distal to the duodeno-jejunal junction. After completion of the resection, the proximal end of the first loop of jejunum was then brought through the transverse mesocolon, and the gastrojejunal anastomosis (GJA) was performed in two layers by using 3-0 PDS sutures and 4-0 silk sutures in an end-to-side fashion. The jejunum was then divided 35 to 40 cm distal to the GJA, and the distal limb was brought separately through the transverse mesocolon to be placed in the duodenal bed for reconstruction of the pancreatojejunal anastomosis (PJA) and hepatojejunal anastomosis (HJA).
  Arms: PrPD with RGA
Procedure: conventional PrPD — After completion of the pancreatojejunal anastomosis (PJA) and hepatojejunal anastomosis (HJA), a hand-sewn, isoperistaltic GJA was performed 25 to 30 cm distal to the HJA in two layers by using 3-0 polydioxanone (PDS) sutures and 4-0 silk sutures.
  Arms: conventional PrPD

SUMMARY:
This study aims to evaluate whether the incidence of delayed gastric emptying (DGE) can be reduced by proximal Roux-en-y gastrojejunal anastomosis in comparison with the standard gastrojejunal anastomosis in pylorus-resecting pancreaticoduodenectomy (PrPD).

DETAILED DESCRIPTION:
Delayed gastric emptying (DGE) is a common complication after pancreaticoduodenectomy (PD), occurring in 20% to 70% of the patients. DGE is usually not a life-threatening complication, but it contributes significantly to increased length of hospital stay, health care costs, and patient discomfort. In a recent study by Sakamoto et al, proximal Roux-en-y gastrojejunal anastomosis is associated with a reduced incidence of DGE after pylorus-resecting pancreaticoduodenectomy (PrPD); however, these results may have been biased because of the retrospective nature. Therefore, the investigators conducted the present randomized controlled trial (RCT) to evaluate the impact of the proximal Roux-en-y gastrojejunal anastomosis on reducing DGE following PrPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled to undergo PD and provided written informed consent.
* In the opinion of the surgeon, the subject has no medical contraindications to PD.
* At least 18 years of age.

Exclusion Criteria:

* Patients who underwent other surgical procedures than PD, such as total pancreatectomy (TP) or a palliative biliary and gastroenteric anastomosis.
* Drug abusers or alcoholics.
* Patient who have previous transabdominal surgery.
* The patient who were scheduled to undergo laparoscopic PD.
* The patient who does not want to participate the clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Delayed gastric emptying,rate | 60 days after operation
  The severity of DGE was classified into 3 grades (A, B, or C) according to the ISGPS's clinical criteria, based on the patient's clinical course and postoperative management, such as the need for NGT in the postoperative period or the inability to tolerate solid oral intake.
  Grade A was defined as needing the NGT for more than 7 days or reinsertion of the NGT after postoperative day 3, or as being unable to tolerate a solid diet by postoperative day 7.
  Grade B was defined as needing for NGT for 8 to 14 days after surgery or reinsertion of the NGT after day 7, or as being unable to tolerate a solid diet by postoperative day 14.
  Grade C was defined as needing the NGT for more than 14 days or reinsertion of the NGT after day 14, or as being unable to tolerate a solid diet by day 21.

SECONDARY OUTCOMES:
Morbidity,rate | 60 days after operation
Mortality,rate | 60 days after operation
Length of hospital stay,days | 60 days after operation
Pancreatic fistula,rate | 60 days after operation
Hemorrhage,rate | 60 days after operation
Bile leakage,rate | 60 days after operation
Intra-abdominal abscess,rate | 60 days after operation
wound infection,rate | 60 days after operation

OTHER OUTCOMES:
nonsurgical complications,rate | 60 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Zhou, Dr, Principal Investigator — First affiliated Hospital of Xiamen University
Locations (1):
- First affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data.

REFERENCES:
- [Result] Barakat O, Cagigas MN, Bozorgui S, Ozaki CF, Wood RP. Proximal Roux-en-y Gastrojejunal Anastomosis with Pyloric Ring Resection Improves Gastric Emptying After Pancreaticoduodenectomy. J Gastrointest Surg. 2016 May;20(5):914-23. doi: 10.1007/s11605-016-3091-5. Epub 2016 Feb 5. PMID 26850262